CLINICAL TRIAL: NCT04299828
Title: Evaluation of Pro-Inflammatory Leukocyte Activity in Patients Undergoing Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Koichi Yuki, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: P00033314
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease; Coagulation
MeSH Terms: conditions — Heart Defects, Congenital; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Discarded blood samples — Will utilize the discarded blood from routine clinical blood samples to evaluate the role of immune cells in coagulopathy.

SUMMARY:
The goal of this proposal is to prospectively collect data from a series of 200 patients (all ages) undergoing complex cardiac surgical procedures involving cardiopulmonary bypass (CPB) to:

1. Measure the number of blood activated circulating monocytes before, during and after cardiac surgery and serum GABA and pro-inflammatory cytokine levels
2. Understand the correlation between GABA and inflammatory cytokines (and/or activated monocytes) and
3. Assess the correlation between thrombosis and monocyte activation in patients undergoing cardiac surgery under CPB and at risk of thrombosis.

DETAILED DESCRIPTION:
Often when people undergo heart surgery, they are placed on cardiopulmonary bypass (CPB). Sometimes clotting of the blood occurs during and after heart surgery with CPB, which can lead to multiple complications. In order to try to avoid abnormal/excessive clotting that may lead to complications, it is important to understand the specific causes of why the blood sometimes clots abnormally during and after heart surgery.

Currently, tests looking at how the blood clots (coagulation assessment) are usually performed as standard laboratory testing during and after surgery. However, these tests are not able to predict the future development of abnormal clots.

This study will be looking at the role that immune cells (monocytes) have in the formation of abnormal clots after heart surgery. It is possible that these immune cells produce signals that can contribute to the formation of clots. Using experimental tests (monocyte analysis and mediator analysis), the hope is to understand if these cells participate in forming abnormal clots in any meaningful way. Although these tests are not yet approved for use in children, this study plans to use these new methods to understand this phenomenon by analyzing the blood at different times during the surgery and recovery period.

Overall, the purpose of this study is to look at these tests in people undergoing heart surgery to help the investigators understand why the blood sometimes forms clots abnormally. Results from this study may help treat future patients who experience abnormal clotting during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients (all ages) undergoing complex cardiac surgical procedures with CPB.

Exclusion Criteria:

* undergoing an emergent procedure and do not have more than 1 hour ahead of time to review the consent
* patient in a moribund condition American Society of Anesthesiology (ASA 5) -patient with a hematological and/or oncological disease
* Jehovah witnesses.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (all ages) undergoing complex cardiac surgical procedures with cardiopulmonary bypass (CPB) at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Monocyte activation status | Through study completion; on average one year
  characterization of monocyte activation status at baseline before surgery and throughout the course of CPB including post-operatively.
Serum GABA and pro-inflammatory cytokines | Through study completion; on average one year
  Serum GABA and pro-inflammatory cytokines

SECONDARY OUTCOMES:
Clinical Thrombosis | Through study completion; on average one year
  Presence of clinical thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Yuki, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No